CLINICAL TRIAL: NCT00854165
Title: Extracorporeal Membrane Oxygenation Support for Bilateral Sequential Lung Transplantation in Respiratory Failure Patients.
Brief Title: Lung Transplantation in Respiratory Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yung-Chie Lee, Department of Surgery
Other Study IDs: 200901015R
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Respiratory Failure
Keywords: lung transplantation; respiratory failure; ECMO; Lung transplants in respiratory failure patients
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Survival after cadaveric lung transplantation in recipients depended on ventilation support prior to transplantation has been reported to have relative high surgical mortality and morbidity rate. The objectives of this study were to describe the short-term outcomes of bilateral sequential lung transplantation under extracorporeal membrane oxygenation (ECMO) support in a consecutive series of patients who depended on noninvasive and invasive ventilation support preoperatively .

DETAILED DESCRIPTION:
The one-year survival rate and postoperative pulmonary functional results will be reported in this study.

ELIGIBILITY:
Inclusion Criteria:

* respiratory patients depended on ventilator supports prior to lung transplant

Exclusion Criteria:

* non-cardaveric lung transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between July 2006 and July 2008, we performed bilateral sequential lung transplantation under venoarterious ECMO support in 10 respiratory failure patients with various lung diseases. This study wanted to report the preoperative condition, postoperative complications, and short-term outcome after lung transplantation.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
6 months and one year survival after lung transplatn. | 6 months and one year posttransplant

SECONDARY OUTCOMES:
Pulmonary function results, at baseline and posttransplant 1, 3, and 6 months. | baseline, post-op 1,3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chie Lee, MD, PhD, Study Director — Department of Surgery, National Taiwan University Hospital; Hsao-Hsun Hsu, MD, Principal Investigator — Department of Surgery, National Taiwan University Hospital
Locations (1):
- Department of Surgery, National Taiwan University Hospital, Taipei, Taiwan